CLINICAL TRIAL: NCT03761394
Title: Smartwatch Monitoring for Atrial Fibrillation After Stroke
Brief Title: Pulsewatch: Smartwatch Monitoring for Atrial Fibrillation After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: University of Connecticut (Other); Northeastern University (Other); Brigham and Women's Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Timothy P Fitzgibbons, MD, PhD, Assistant Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: H00016067; R01HL137734-01A1 (NIH)
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Atrial Fibrillation
Keywords: Cardiac Arrhythmias
MeSH Terms: conditions — Stroke; Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Intervention Group (Experimental): Testing devices plus Cardea Solo device by Cardiac Insight for 14-day period.
  Interventions: Device: Testing Devices; Device: Cardea Solo by Cardiac Insight
- Control Group (Active Comparator): Only Cardea Solo device by Cardiac Insight for 14-day period.
  Interventions: Device: Cardea Solo by Cardiac Insight
- Intervention Group for Extended Use (Experimental): 30-additional days of extended use of testing devices for adherence plus Kardia Mobile ECG device by AliveCor.
  Interventions: Device: Testing Devices; Device: Kardia Mobile by AliveCor
- Control Group for Extended Use (No Intervention): No device usage for 30-days following completion of the original 14-day period.

INTERVENTIONS:
Device: Testing Devices — Pulsewatch system testing application on smartphone with smartwatch.
  Arms: Intervention Group; Intervention Group for Extended Use
Device: Cardea Solo by Cardiac Insight — Gold-standard cardiac monitor for comparison of testing devices.
  Arms: Control Group; Intervention Group
Device: Kardia Mobile by AliveCor — Mobile ECG device for comparison of testing devices during the extended use period.
  Arms: Intervention Group for Extended Use

SUMMARY:
The goal of this research study is to develop a smartphone application capable of monitoring paroxysmal atrial fibrillation (pAF) in people who have survived a stroke or transient ischemic attack (TIA) or people who are at risk for a stroke and are age 50 and older. The study team plans to develop a highly effective and easy to use cardiovascular surveillance system to monitor patients for pAF on a nearly continuous basis. People involved in the development of this system include patients, their caregivers, health care providers, and computer programmers.

ELIGIBILITY:
Inclusion Criteria:

* History of Transient Ischemic Attack (TIA) or stroke or at risk for stroke based on a CHA2DS2-VASc score equal to or greater to a score of 3, presenting at the UMass Memorial Medical Center (UMMMC) inpatient service or ambulatory clinic (neurology clinics and cardiovascular clinics included)
* Age: greater to or equal to 50 years of age
* Able to sign informed consent
* Willing to participant in a focus groups and/or Hack-a-thon for Aim 1 participants only
* Willing and capable of using Pulsewatch (smartwatch and smartphone app) daily for up to 44-days and returning to UMMMC for up to two study visits for Aims 2 and 3 participants only

Exclusion Criteria:

* Major contraindication to anti-coagulation treatment
* Plans to move our of the area over the 44-day follow up period
* Serious physical illness (e.g., unable to interact with a smart device, or communicate verbally or via written text) that would interfere with study participation
* Known allergies or hypersensitivities to medical grade hydrocolloid adhesives or hydrogel
* Patient with life threatening arrhythmia's who require in-patient monitoring for immediate analysis
* Patient with implantable pacemaker as paced beats interfere with ECG readings
* Lacking capacity to sign informed consent
* Unable to read and write in English
* Plans to move from the area during the study period
* Unwilling to complete all study procedures
* Major contraindication to anti-coagulation treatment (i.e., major hemorrhagic stroke)
* Individuals who are not yet adults
* Pregnant women
* Prisoners

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Fitzgibbons, MD, PhD, Principal Investigator — UMass Medical School
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ding EY, Tran KV, Lessard D, Wang Z, Han D, Mohagheghian F, Mensah Otabil E, Noorishirazi K, Mehawej J, Filippaios A, Naeem S, Gottbrecht MF, Fitzgibbons TP, Saczynski JS, Barton B, Chon K, McManus DD. Accuracy, Usability, and Adherence of Smartwatches for Atrial Fibrillation Detection in Older Adults After Stroke: Randomized Controlled Trial. JMIR Cardio. 2023 Nov 28;7:e45137. doi: 10.2196/45137. PMID 38015598
- [Derived] Han D, Ding EY, Cho C, Jung H, Dickson EL, Mohagheghian F, Peitzsch AG, DiMezza D, Tran KV, McManus DD, Chon KH. A Smartwatch System for Continuous Monitoring of Atrial Fibrillation in Older Adults After Stroke or Transient Ischemic Attack: Application Design Study. JMIR Cardio. 2023 Feb 13;7:e41691. doi: 10.2196/41691. PMID 36780211

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruitment period was from September 2019 to September 2021. Participants were recruited from neurology and cardiology clinics at UMass Memorial and the Ambulatory Care Center, respectively. After participants were agreeable to joining the study, we gave them an IRB-stamped consent form that detailed the study's protocol. All study staff members were trained properly and had a complete understanding of study-related documentation to help answer any questions participants may have.
Pre-assignment Details: Patients were either randomized into the intervention or control arm of the study. The control patients were given a gold-standard cardiac monitor patch (2 patches over 14 days) but were not offered the use of the Pulsewatch system. Thereafter, we re-randomized the 120 participants into a 1:1 randomization of control group (n=60) and intervention group (n=60) to continue using the device for an additional 30 days. Control group did not receive any devices during this time.
Period: 14-day Intervention & Control Period
Arm/Group | Intervention Group | Control Group | Intervention Group for Extended Use | Control Group for Extended Use
Started | 90 | 30 | 0 | 0
Completed | 87 | 28 | 0 | 0
Not Completed | 3 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 0
Period: 30-day Period (Extension 44 Days)
Arm/Group | Intervention Group | Control Group | Intervention Group for Extended Use | Control Group for Extended Use
Started | 0 | 0 | 57 | 58
Completed | 0 | 0 | 55 | 55
Not Completed | 0 | 0 | 2 | 3
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Participants in the "Intervention Group for Extended Use" and "Control Group for Extended Use" did not complete baseline assessments as they are a continuation of the arms
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Intervention Group for Extended Use | Control Group for Extended Use | Total
Number analyzed (Participants) | 89 | 30 | 0 | 0 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  |  | 0
  Between 18 and 65 years | 35 | 11 |  |  | 46
  >=65 years | 54 | 19 |  |  | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (9.5) | 68.3 (8.68) |  |  | 67.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 13 |  |  | 50
  Male | 52 | 17 |  |  | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 6 |  |  | 20
  Not Hispanic or Latino | 75 | 24 |  |  | 99
  Unknown or Not Reported | 0 | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 |  |  | 2
  Asian | 1 | 1 |  |  | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
  Black or African American | 5 | 0 |  |  | 5
  White | 77 | 26 |  |  | 103
  More than one race | 2 | 1 |  |  | 3
  Unknown or Not Reported | 3 | 1 |  |  | 4
Region of Enrollment [Number; unit: participants]
  United States | 89 | 30 |  |  | 119

OUTCOME MEASURES:

1. Primary Outcome: Usability of Pulsewatch System (System Usability Scale & Rating Scale) at 14 Days Post the First Randomization
Description: System usability scale, self-reported, of likes, dislikes, and problems encountered with the smartphone application and smartwatch. Each item regarding likes and dislikes will be scored 1-5 (1= strongly disagree; 5= strongly agree or Didn't use). Problem encountered will be scored with yes or no options with space provided for explanations. Also, using Mobile Application Rating Scale (MARS) App Classification questions will capture the participants' experience with the application. Each MARS item uses a 5-point scale (1=inadequate, 2=poor, 3=acceptable, 4=Good, 5=Excellent) and sub-scales will have an average mean to indicate the overall rating of the application.
  Number of participants with SUS > 68 was reported in the Outcome Measure Data Table
Time Frame: Assessed 14 days post the first randomization
Population: Only the intervention group in the first phase had outcomes assessed for their Pulsewatch system usability. The overall number analyzed is 83 instead of 90 because 3 participants withdrew and the other 4 participants either had their device lost in transit or the data was not able to sync.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group | Intervention Group for Extended Use | Control Group for Extended Use
Number analyzed (Participants) | 83 | 0 | 0 | 0
Participants | 31 |  |  |

2. Primary Outcome: The Number of Participants With Atrial Fibrillation Detected by Smartwatch at the 14 Day Trial Period
Description: This outcome was measured by the number of atrial fibrillation episodes identified by the smartwatch biosensors. This was conducted using two approaches. Firstly, the Pulsewatch app sent a message to participants to remain still and perform a 30-sec ECG self-check (wrist electrode, high accuracy) should they have an AF episode detected. The second approach involved the cancellation of cyclical frequencies, seen in accelerometer data, from the photoplethysmogram (PPG) signal. Thus, these two approaches were effectively used to recover some data segments contaminated by MNA or by poor signal quality and correctly identified the presence or absence of AF. Once MN artifacts were corrected, we looked at patterns to analyze pulse waveforms for AF detection, including discrimination of PVCs and PACs
Time Frame: Assessed throughout 14 day trial period
Population: Control, Intervention Group for Extended Use, and Control Group for Extended Use Groups analyses are not applicable. The number of participants analyzed is 89 because one participant's device was lost in transit so we were unable to get the device to extract the data.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group | Intervention Group for Extended Use | Control Group for Extended Use
Number analyzed (Participants) | 89 | 0 | 0 | 0
Participants | 7 |  |  |

3. Primary Outcome: The Number of Participants With Detection of Atrial Fibrillation by a Patch Monitor (Confirmed by Cardiologist Overread) at 14 Days Post the First Randomization.
Description: Episodes of atrial fibrillation was identified by the gold-standard monitor (Cardea Solo by Cardiac Insight). The Cardiac Insight patches have a module chip inside the sensor that stores the data being collected over the 14-days. After the participants returned the patches at the end of the 14-day monitoring period, a trained study staff removed the modules and placed them into the Cardiac insight smart cable to be uploaded to a UMass Medical School server. The ECG readings are then read by a board-certified cardiologist to confirm true atrial fibrillation detection.
Time Frame: Assessed at 14 days post the first randomization.
Population: Intervention Group for Extended Use and Control Group for Extended Use analyses are not applicable. One participant did not activate their Cardea solo device and one participant could discontinued wearing the device due to allergic reaction.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group | Intervention Group for Extended Use | Control Group for Extended Use
Number analyzed (Participants) | 88 | 29 | 0 | 0
Participants | 6 | 0 |  |

4. Secondary Outcome: Change in Anxiety Symptoms at Baseline and at the Last Study Visit 30 Days Post the Second Randomization.
Description: Anxiety will be assessed using the Generalized Anxiety Disorder-7 scale (GAD-7), a revised version of the anxiety module from the Patient Health Questionnaire, which consists of Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for generalized anxiety disorder over the past 2 weeks. The GAD-7 score ranges from 0-27 with scores of 5, 10 and 15 representing validated cut-points for mild, moderate and severe levels of anxiety symptoms, with a score ≥10 having high sensitivity (0.89) and specificity (0.82) for psychiatrist diagnosed anxiety disorder and correlates significantly with health-related QoL. This change in outcome was between baseline and the last study visit 30 days post the second randomization.
Time Frame: Assessed at baseline and at the last study visit 30 days post the second randomization (44 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group | Intervention Group for Extended Use | Control Group for Extended Use
Number analyzed (Participants) | 41 | 13 | 41 | 13
score on a scale | 0.17 (3.61) | -0.77 (2.39) | 0.56 (3.44) | -0.46 (3.69)

5. Secondary Outcome: Change in General Health MCS at Baseline and at the Last Study Visit 30 Days Post the Second Randomization (44 Days)
Description: The Short Form (SF-12) health survey to assess health related quality of life, this validated instrument domains include general health questions and mental health related questions. Scores range from 0 to 100, where higher scores indicate higher level of health. This change in outcome was between baseline and the last study visit 30 days post the second randomization (44 days).
Time Frame: Assessed at baseline and at the last study visit 30 days post the second randomization (44 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group | Intervention Group for Extended Use | Control Group for Extended Use
Number analyzed (Participants) | 41 | 14 | 41 | 13
score on a scale | 1.56 (6.79) | 3.10 (6.29) | 2.90 (7.51) | 1.08 (6.38)

6. Secondary Outcome: Change in General Health PCS at Baseline and at the Last Study Visit 30 Days Post the Second Randomization (44 Days)
Description: The Short Form (SF-12) health survey to assess health related quality of life, this validated instrument domains include general health questions and physical health-related questions. Scores range from 0 to 100, where higher scores indicate a higher level of health. This outcome was assessed at baseline and at the last study visit 30 days post the second randomization (44 days).
Time Frame: Assessed at baseline and at the last study visit 30 days post the second randomization (44 days)
Population: The outcome measure timeframe is at baseline and at the last study visit 30 days post the second randomization (44 days) for both control and intervention groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group | Intervention Group for Extended Use | Control Group for Extended Use
Number analyzed (Participants) | 41 | 14 | 41 | 13
score on a scale | 0.35 (6.86) | 0.27 (3.42) | -0.04 (6.03) | 0.36 (4.60)

7. Secondary Outcome: Change in Disease Management Self-Efficacy (The General Disease Management Scale) at Baseline and 14 Days Post the First Randomization
Description: Self-efficacy for disease management is associated with engagement in health behaviors and with improved medication adherence. The General Disease Management scale is a 5-item scale assessing confidence in disease self-management (scores 0-50, higher scores = greater confidence, lower scores = lower confidence). This change in outcome was between baseline and 14 days post the first randomization.
Time Frame: Assessed at baseline and 14 days post the first randomization
Population: The outcome measure timeframe is at baseline and 14 days post-randomization. Intervention Group for Extended Use and Control Group for Extended Use are not applicable to this analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group | Intervention Group for Extended Use | Control Group for Extended Use
Number analyzed (Participants) | 82 | 27 | 0 | 0
score on a scale | 0.67 (5.76) | -9.03 (4.79) |  |

8. Secondary Outcome: Change in Symptom Management Self-Efficacy at Baseline and 14 Days Post Randomization
Description: Self-efficacy for disease management is associated with engagement in health behaviors and with improved medication adherence. The Symptom Management scale is a 5-item scale assessing confidence in managing chronic disease symptoms (items tailored to the sample), with scores ranging from 0 to 100. A higher symptom management score indicates a higher confidence in managing symptoms. Conversely, a lower score indicates a lower confidence in managing symptoms. This change in outcome was between baseline and 14 days post randomization.
Time Frame: Assessed at baseline and 14 days post randomization
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group | Intervention Group for Extended Use | Control Group for Extended Use
Number analyzed (Participants) | 82 | 27 | 0 | 0
score on a scale | 1.52 (8.81) | 0.74 (4.61) |  |

9. Secondary Outcome: Change in Patient Activation Score at Baseline and at the Last Study Visit 30 Days Post the Second Randomization (44 Days)
Description: Patient activation refers to a patient's ability and willingness to manage their health. Activation will be measured using the 10-item Consumer Health Activation Index (CHAI). Scores range from 10 to 60. A higher score indicates that the patient has higher activation for self-management of their condition. Conversely, a lower score indicates lower activation for self-management of their condition. This change in outcome was between the baseline and the last study visit 30 days post the second randomization (44 days)
Time Frame: Assessed at baseline and at the last study visit 30 days post the second randomization (44 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group | Intervention Group for Extended Use | Control Group for Extended Use
Number analyzed (Participants) | 40 | 14 | 41 | 13
score on a scale | 3.75 (15.35) | 2.00 (5.71) | 4.29 (10.57) | 1.54 (6.98)

10. Secondary Outcome: Change in Medication Adherence at Baseline and 14 Days Post the First Randomization
Description: Medication adherence will be measured using the 12-item Adherence to Refills and Medications Scale (ARMS), a well-validated measure of patient-reported adherence. The minimum to maximum ARMS score ranges from 1 to 4. Higher scores indicate poorer adherence, and lower scores indicate better medication adherence. This change in outcome was between baseline and 14 days post the first randomization.
Time Frame: Assessed at baseline and 14 days post the first randomization
Population: Only the intervention group has analyzable data for this outcome. Control Group, Intervention Group for Extended Use, and Control Group for Extended Use are not applicable to this analysis. The number of participants analyzed was 76 because participants either withdrew, were lost to follow-up, or skipped these questions on the questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group | Intervention Group for Extended Use | Control Group for Extended Use
Number analyzed (Participants) | 76 | 0 | 0 | 0
score on a scale | -1.12 (2.50) |  |  |

ADVERSE EVENTS:
Time Frame: The adverse event data were monitored at baseline, at 14 days, and the 30 additional day follow-up for a total of approximately 44 days. Patient 1 - Serious adverse event occurred during the 14-day period. Patient 2 - Serious adverse event occurred during the 14-day period. Patient 3 - Serious adverse event occurred during the 14-day period. Patient 4 - Serious adverse event occurred during the 30-day extended period.
Description: The definition of adverse event and/or serious adverse event used in this study was adapted from the clinicaltrials.gov definitions.
  The study principal investigator and data safety monitor were promptly notified of all adverse and serious adverse events and were asked for guidance on what action should be taken.
  All adverse events and serious adverse events were recorded in REDCap, a data collection tool, and also to the UMass Chan IRB
Arm/Group | Intervention Group | Control Group | Intervention Group for Extended Use | Control Group for Extended Use
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/30 | 0/57 | 0/58
Serious Adverse Events (participants affected / at risk) | 1/90 | 2/30 | 1/57 | 0/58
Other Adverse Events (participants affected / at risk) | 1/90 | 3/30 | 0/57 | 0/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=90) | Control Group (N=30) | Intervention Group for Extended Use (N=57) | Control Group for Extended Use (N=58)
Myocardial infarction and hospitalization (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | NA — The patient had a myocardial infarction and was hospitalized for a period of time. This was completely unrelated to our study protocol/procedures. Once the patient was discharged, they withdrew and wanted to focus on recovering from the event.
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | NA — The participant was admitted to the hospital on 3/27/2020 with weakness and a nonproductive cough. He was diagnosed with a COVID-19 infection. He was then discharged on 3/28/2020 with instructions to self-quarantine
Chest Pain and hospitalization (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | NA — The patient was hospitalized for chest pain on 6/10/2021
Pancreatitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | NA — The patient was hospitalized for pancreatitis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=90) | Control Group (N=30) | Intervention Group for Extended Use (N=57) | Control Group for Extended Use (N=58)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | NA | NA — Participants had skin irritation to the Cardiac Insight patch. They were asked to remove the Cardiac Insight patch and not place their second patch.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/94/NCT03761394/Prot_008.pdf
  • Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT03761394/SAP_003.pdf